CLINICAL TRIAL: NCT03949127
Title: Efficacy of a Non-surgical Treatment Protocol for Patients With Symptomatic Femoro-acetabular Impingement: a Randomized Controlled Trial
Brief Title: Efficacy of an Exercise Program for Patients With Femoro-acetabular Impingement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Orthopaedic Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20190091
Record Dates: First submitted 2019-04-14; First posted 2019-05-14 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Femoracetabular Impingement
Keywords: non-surgical treatment; exercise
MeSH Terms: conditions — Femoracetabular Impingement; Motor Activity

STUDY DESIGN:
Intervention Model Description: There will be two groups, one will be the exercise group and one will be used as a control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): The group who will exercise to manage pain.
  Interventions: Other: Exercise Group
- Control Group (No Intervention): The group who will not take part in any exercises and only have to do assessments.

INTERVENTIONS:
Other: Exercise Group — The group who will meet a physiotherapist who will show them strengthening and stretching muscles associated with pelvic tilt.
  Arms: Exercise Group

SUMMARY:
The purpose of this study is to examine whether using an exercise regime on people with femoroacetabular impingement (FAI) can help reduce pain and improve function. Also, it examines whether the exercise regime will help prevent the worsening of hip cartilage deterioration.

DETAILED DESCRIPTION:
A significant proportion of adults from ages 18 to 50 have a deformity in the neck of their femur. This can be painful and is called a femoroacetabular impingement (FAI), and could lead to ones cartilage being destroyed and possibly lead to osteoarthritis of the hip. People with this deformity in their femur have been found to move their hips differently when doing tasks such as walking, squatting or climbing stairs compared to those without this problem. The investigators are testing whether exercise that targets this difference in movement can help reduce pain, improve function and prevent cartilage damage. There will recruit 84 patients with divided into 2 groups. 42 patients will do a 8 week exercise program on strengthening muscles responsible for extending the hip and stretching muscles that are associated with flexing the hip. The intensity of the program will change with visits to the physiotherapist through the course of their exercise program. This research hopes to develop an innovative, non-surgical, low-cost, highly feasible and accessible intervention for patients with FAI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with symptomatic FAI
* at least 3 months of groin pain
* increased pain with hip rotation
* an alpha angle greater than 60 degrees on multiplane imaging
* labral tear on MRI
* Tonnis grade of 0 or 1

Exclusion Criteria:

* diagnosed health problems other than FAI interfering with capacity to accomplish the exercise program
* previous hip surgery on the affected side
* surgery will happen within 6 months

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Estimated)
Dates: Start 2019-09-06 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
iHOT-33 | Change in Baseline before exercise program and 6 months
  International Hip Outcome Tool-33, disease-specific function. Each answer will be measured on a scale of 100mm and the mean of the 33 questions will be taken as a final score. A higher score indicates a better quality of life.

SECONDARY OUTCOMES:
EQ-5D-5L | Change in Baseline before exercise program and 6 months afterward
  Generic quality of life, the scores for each question are summed up for a total with a higher score being a better quality of life.
Number of participants that receive hip surgery | Change in Baseline before exercise program and 1 year afterwards
  If the participant has hip surgery in the time frame
Patient-reported hip pain | Change in Baseline before exercise program and 6 months
  Patient perceived pain on a VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Paul Beaule, MD, FRCSC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khanna V, Beaule PE. Defining structural abnormalities of the hip joint at risk of degeneration. J Hip Preserv Surg. 2014 Sep 6;1(1):12-20. doi: 10.1093/jhps/hnu004. eCollection 2014 Jul. PMID 27011797
- [Background] Khanna V, Caragianis A, Diprimio G, Rakhra K, Beaule PE. Incidence of hip pain in a prospective cohort of asymptomatic volunteers: is the cam deformity a risk factor for hip pain? Am J Sports Med. 2014 Apr;42(4):793-7. doi: 10.1177/0363546513518417. Epub 2014 Jan 30. PMID 24481825
- [Background] Diamond LE, Dobson FL, Bennell KL, Wrigley TV, Hodges PW, Hinman RS. Physical impairments and activity limitations in people with femoroacetabular impingement: a systematic review. Br J Sports Med. 2015 Feb;49(4):230-42. doi: 10.1136/bjsports-2013-093340. Epub 2014 Sep 22. PMID 25246442
- [Background] Hack K, Di Primio G, Rakhra K, Beaule PE. Prevalence of cam-type femoroacetabular impingement morphology in asymptomatic volunteers. J Bone Joint Surg Am. 2010 Oct 20;92(14):2436-44. doi: 10.2106/JBJS.J.01280. PMID 20962194
- [Background] Peters CL. Mild to Moderate Hip OA: Joint Preservation or Total Hip Arthroplasty? J Arthroplasty. 2015 Jul;30(7):1109-12. doi: 10.1016/j.arth.2015.02.046. Epub 2015 Mar 25. PMID 25842248
- [Background] Beaule PE, Singh A, Poitras S, Parker G. Surgical Dislocation of the Hip for the Treatment of Pre-Arthritic Hip Disease. J Arthroplasty. 2015 Sep;30(9):1502-5. doi: 10.1016/j.arth.2015.04.009. Epub 2015 Apr 11. PMID 25913231
- [Background] Speirs AD, Beaule PE, Rakhra KS, Schweitzer ME, Frei H. Increased acetabular subchondral bone density is associated with cam-type femoroacetabular impingement. Osteoarthritis Cartilage. 2013 Apr;21(4):551-8. doi: 10.1016/j.joca.2013.01.012. Epub 2013 Jan 26. PMID 23357224
- [Background] Speirs AD, Beaule PE, Huang A, Frei H. Properties of the cartilage layer from the cam-type hip impingement deformity. J Biomech. 2017 Apr 11;55:78-84. doi: 10.1016/j.jbiomech.2017.02.007. Epub 2017 Feb 21. PMID 28259463
- [Background] Carsen S, Moroz PJ, Rakhra K, Ward LM, Dunlap H, Hay JA, Willis RB, Beaule PE. The Otto Aufranc Award. On the etiology of the cam deformity: a cross-sectional pediatric MRI study. Clin Orthop Relat Res. 2014 Feb;472(2):430-6. doi: 10.1007/s11999-013-2990-y. PMID 23604603
- [Background] Gala L, Khanna V, Rakhra KS, Beaule PE. Does the femoral head/neck contour in the skeletally mature change over time? J Hip Preserv Surg. 2016 Aug 3;3(4):333-337. doi: 10.1093/jhps/hnw022. eCollection 2016 Oct. PMID 29632694
- [Background] Li X, Majumdar S. Quantitative MRI of articular cartilage and its clinical applications. J Magn Reson Imaging. 2013 Nov;38(5):991-1008. doi: 10.1002/jmri.24313. Epub 2013 Oct 2. PMID 24115571
- [Background] Anwander H, Melkus G, Rakhra KS, Beaule PE. T1rho MRI detects cartilage damage in asymptomatic individuals with a cam deformity. J Orthop Res. 2016 Jun;34(6):1004-9. doi: 10.1002/jor.23101. Epub 2015 Dec 2. PMID 26573964
- [Background] Beaule PE, Speirs AD, Anwander H, Melkus G, Rakhra K, Frei H, Lamontagne M. Surgical Correction of Cam Deformity in Association with Femoroacetabular Impingement and Its Impact on the Degenerative Process within the Hip Joint. J Bone Joint Surg Am. 2017 Aug 16;99(16):1373-1381. doi: 10.2106/JBJS.16.00415. PMID 28816897
- [Background] Fairley J, Wang Y, Teichtahl AJ, Seneviwickrama M, Wluka AE, Brady SRE, Hussain SM, Liew S, Cicuttini FM. Management options for femoroacetabular impingement: a systematic review of symptom and structural outcomes. Osteoarthritis Cartilage. 2016 Oct;24(10):1682-1696. doi: 10.1016/j.joca.2016.04.014. Epub 2016 Apr 20. PMID 27107630
- [Background] Wall PD, Fernandez M, Griffin DR, Foster NE. Nonoperative treatment for femoroacetabular impingement: a systematic review of the literature. PM R. 2013 May;5(5):418-26. doi: 10.1016/j.pmrj.2013.02.005. Epub 2013 Feb 16. PMID 23419746
- [Background] Lamontagne M, Kennedy MJ, Beaule PE. The effect of cam FAI on hip and pelvic motion during maximum squat. Clin Orthop Relat Res. 2009 Mar;467(3):645-50. doi: 10.1007/s11999-008-0620-x. Epub 2008 Nov 26. PMID 19034598
- [Background] Seijas R, Alentorn-Geli E, Alvarez-Diaz P, Marin M, Ares O, Sallent A, Cusco X, Cugat R. Gluteus maximus impairment in femoroacetabular impingement: a tensiomyographic evaluation of a clinical fact. Arch Orthop Trauma Surg. 2016 Jun;136(6):785-9. doi: 10.1007/s00402-016-2428-6. Epub 2016 Feb 25. PMID 26914331
- [Background] Ross JR, Nepple JJ, Philippon MJ, Kelly BT, Larson CM, Bedi A. Effect of changes in pelvic tilt on range of motion to impingement and radiographic parameters of acetabular morphologic characteristics. Am J Sports Med. 2014 Oct;42(10):2402-9. doi: 10.1177/0363546514541229. Epub 2014 Jul 24. PMID 25060073
- [Background] Nepple JJ, Prather H, Trousdale RT, Clohisy JC, Beaule PE, Glyn-Jones S, Kim YJ. Clinical diagnosis of femoroacetabular impingement. J Am Acad Orthop Surg. 2013;21 Suppl 1:S16-9. doi: 10.5435/JAAOS-21-07-S16. PMID 23818186
- [Background] Nwachukwu BU, Fields K, Chang B, Nawabi DH, Kelly BT, Ranawat AS. Preoperative Outcome Scores Are Predictive of Achieving the Minimal Clinically Important Difference After Arthroscopic Treatment of Femoroacetabular Impingement. Am J Sports Med. 2017 Mar;45(3):612-619. doi: 10.1177/0363546516669325. Epub 2016 Oct 23. PMID 27765733
- [Background] Wright AA, Hegedus EJ, Taylor JB, Dischiavi SL, Stubbs AJ. Non-operative management of femoroacetabular impingement: A prospective, randomized controlled clinical trial pilot study. J Sci Med Sport. 2016 Sep;19(9):716-21. doi: 10.1016/j.jsams.2015.11.008. Epub 2016 Jan 6. PMID 26795448
- [Background] Coppack RJ, Bilzon JL, Wills AK, McCurdie IM, Partridge LK, Nicol AM, Bennett AN. Physical and functional outcomes following multidisciplinary residential rehabilitation for prearthritic hip pain among young active UK military personnel. BMJ Open Sport Exerc Med. 2016 Apr 1;2(1):e000107. doi: 10.1136/bmjsem-2015-000107. eCollection 2016. PMID 27900174
- [Background] Griffin D, Wall P, Realpe A, Adams A, Parsons N, Hobson R, Achten J, Fry J, Costa M, Petrou S, Foster N, Donovan J. UK FASHIoN: feasibility study of a randomised controlled trial of arthroscopic surgery for hip impingement compared with best conservative care. Health Technol Assess. 2016 Apr;20(32):1-172. doi: 10.3310/hta20320. PMID 27117505
- [Background] Crawford MJ, Dy CJ, Alexander JW, Thompson M, Schroder SJ, Vega CE, Patel RV, Miller AR, McCarthy JC, Lowe WR, Noble PC. The 2007 Frank Stinchfield Award. The biomechanics of the hip labrum and the stability of the hip. Clin Orthop Relat Res. 2007 Dec;465:16-22. doi: 10.1097/BLO.0b013e31815b181f. PMID 17906586
- [Background] Kapron AL, Aoki SK, Peters CL, Anderson AE. Subject-specific patterns of femur-labrum contact are complex and vary in asymptomatic hips and hips with femoroacetabular impingement. Clin Orthop Relat Res. 2014 Dec;472(12):3912-22. doi: 10.1007/s11999-014-3919-9. Epub 2014 Sep 6. PMID 25193693
- [Background] Savic D, Pedoia V, Seo Y, Yang J, Bucknor M, Franc BL, Majumdar S. Imaging Bone-Cartilage Interactions in Osteoarthritis Using [18F]-NaF PET-MRI. Mol Imaging. 2016 Jan 1;15:1-12. doi: 10.1177/1536012116683597. PMID 28654417
- [Background] Pierannunzii L. Pelvic posture and kinematics in femoroacetabular impingement: a systematic review. J Orthop Traumatol. 2017 Sep;18(3):187-196. doi: 10.1007/s10195-016-0439-2. Epub 2017 Feb 1. PMID 28150180